CLINICAL TRIAL: NCT01052779
Title: Ferumoxytol Compared to Iron Sucrose Trial (FIRST): A Randomized, Multicenter, Trial of Ferumoxytol Compared to Iron Sucrose for the Treatment of Iron Deficiency Anemia in Adult Subjects With Chronic Kidney Disease
Brief Title: A Trial Comparing Ferumoxytol to Iron Sucrose for the Treatment of Iron Deficiency Anemia in Adult Subjects With Chronic Kidney Disease
Acronym: FIRST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER-CKD-201; 2009-015630-30 (EudraCT Number)
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Iron Deficiency; Anemia; Kidney Disease
Keywords: Iron deficiency anemia; Chronic kidney disease; Feraheme; Ferumoxytol; Iron sucrose; IDA; CKD; Venofer
MeSH Terms: conditions — Iron Deficiencies; Anemia; Kidney Diseases; Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — Ferrosoferric Oxide; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferumoxytol (Experimental): Participants received an IV injection of ferumoxytol (510 milligrams [mg], 17 milliliters [mL]) on Day 1 (Baseline). This was followed by a second injection of ferumoxytol (510 mg, 17 mL) 5±3 days later for a total cumulative dose of 1.02 grams (g).
  Interventions: Drug: Ferumoxytol
- Iron Sucrose (Active Comparator): Participants received iron sucrose based on hemodialysis status. Participants on hemodialysis received either slow IV injection or IV drip infusion of 100 mg of iron sucrose on Day 1 (Baseline) and at the following 9 consecutive hemodialysis sessions for a total cumulative dose of 1.0 g.
  Participants not on dialysis received either slow IV injection or IV drip infusion of 200 mg of iron sucrose on Day 1 (Baseline) and at 4 subsequent visits on nonconsecutive days over a 14-day period for a total cumulative dose of 1.0 g.
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: Iron Sucrose — IV Iron Sucrose
  Other Names: Venofer
  Arms: Iron Sucrose

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of intravenous (IV) ferumoxytol compared to IV iron sucrose for the treatment of iron deficiency anemia (IDA) in participants with chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria include:

1. Males and females ≥18 years of age
2. An estimated glomerular filtration rate <60 mL/minute or a diagnosis of CKD (such as nephropathy, nephritis)
3. Hemoglobin <11.0 g/deciliter (dL)
4. Transferrin saturation <30%
5. Hemodialysis participants on maintenance dialysis for at least 3 months prior to screening and currently receiving dialysis 3 times per week
6. Female participants of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to screening and agree to remain on birth control until completion of the study

Exclusion Criteria:

Key Exclusion Criteria include:

1. History of allergy to IV iron
2. Allergy to 2 or more classes of drugs
3. Female participants who are pregnant or intend to become pregnant, breastfeeding, within 3 months postpartum, or have a positive serum or urine pregnancy test
4. Hemoglobin ≤7.0 g/dL
5. Received another investigational agent within 4 weeks prior to screening, or planned receipt of an unspecified investigational agent during the study period
6. Known causes of anemia other than iron deficiency (such as hemolysis and vitamin B12 or folate deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2011-07-19 (Actual); Study Completion 2012-04-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tempe, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chula Vista, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mountain View, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meridian, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evergreen Park, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Flushing, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosedale, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Antwerp, Belgium
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond Hill, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Düsseldorf
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Munich
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Passau
- India (3):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangalore
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagpur
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pune
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Opole
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Radom
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- For additional information regarding investigative sites for this trial, contact 1-617-498-3300 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

REFERENCES:
- [Background] Hetzel D, Strauss W, Bernard K, Li Z, Urboniene A, Allen LF. A Phase III, randomized, open-label trial of ferumoxytol compared with iron sucrose for the treatment of iron deficiency anemia in patients with a history of unsatisfactory oral iron therapy. Am J Hematol. 2014 Jun;89(6):646-50. doi: 10.1002/ajh.23712. PMID 24639149
- [Background] Strauss WE, Dahl NV, Li Z, Lau G, Allen LF. Ferumoxytol versus iron sucrose treatment: a post-hoc analysis of randomized controlled trials in patients with varying renal function and iron deficiency anemia. BMC Hematol. 2016 Jul 26;16:20. doi: 10.1186/s12878-016-0060-x. eCollection 2016. PMID 27462400
- [Derived] Macdougall IC, Strauss WE, McLaughlin J, Li Z, Dellanna F, Hertel J. A randomized comparison of ferumoxytol and iron sucrose for treating iron deficiency anemia in patients with CKD. Clin J Am Soc Nephrol. 2014 Apr;9(4):705-12. doi: 10.2215/CJN.05320513. Epub 2014 Jan 23. PMID 24458078

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferumoxytol: Participants received an intravenous (IV) injection of ferumoxytol (510 milligrams [mg], 17 milliliters [mL]) on Day 1 (Baseline). This was followed by a second injection of ferumoxytol (510 mg, 17 mL) 5±3 days later for a total cumulative dose of 1.02 grams (g).
Period: Overall Study
Arm/Group | Ferumoxytol | Iron Sucrose
Started | 80 | 82
Received at Least 1 Dose of Study Drug | 80 | 81
Completed | 75 | 73
Not Completed | 5 | 9
Not completed — Adverse Event | 1 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Other-Protocol Violation | 1 | 1
Not completed — Other-Surgery | 0 | 2
Not completed — Other-Missed Week 5 Visit | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: Any randomized participant who had any exposure to study drug (IV ferumoxytol or IV iron sucrose).
Groups:
- Ferumoxytol: Participants received an IV injection of ferumoxytol (510 mg, 17 mL) on Day 1 (Baseline). This was followed by a second injection of ferumoxytol (510 mg, 17 mL) 5±3 days later for a total cumulative dose of 1.02 g.
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Iron Sucrose | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (15.00) | 63.3 (15.16) | 62.6 (15.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 39 | 80
  Male | 39 | 43 | 82
Dialysis Status [Count of Participants; unit: Participants]
  Hemodialysis | 34 | 36 | 70
  Nondialysis | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Mean Change In Hemoglobin From Baseline (Day 1) To Week 5
Description: The change in hemoglobin from Baseline (Day 1) to Week 5 was calculated for each participant as:
  Hemoglobin Change = Hemoglobin (Week 5) - Hemoglobin (Baseline)
  The least squares mean, with standard error, is reported as g/deciliter (dL). Baseline hemoglobin for each participant was the Day 1 hemoglobin value (prior to injection of the study drug). The screening hemoglobin value was used for any participants with missing Baseline (Day 1) hemoglobin. Analysis used last observed carried forward (LOCF) imputation methods for missing values for the ITT population. Sensitivity analyses were performed without imputation for missing data and with the Markov chain Monte Carlo method.
Time Frame: Baseline (Day 1), Week 5
Population: ITT Population: Any randomized participant who had any exposure to study drug (IV ferumoxytol or IV iron sucrose).
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 80 | 82
g/dL
  With LOCF Imputation | 0.84 (0.14) | 0.74 (0.14)
  Without Imputation (Sensitivity Analysis) | 0.89 (0.15) | 0.80 (0.15)
Statistical Analysis 1: Comparison: Ferumoxytol vs Iron Sucrose; With LOCF Imputation: The p-value and two-sided 95% confidence interval (CI) for the treatment difference in mean change in hemoglobin from Baseline (Day 1) to Week 5 were generated based on an analysis of variance (ANOVA) model adjusted for baseline hemoglobin level and hemodialysis status; Test type: Non-Inferiority — Non-inferiority was concluded if the lower bound of the 95% CI was ≥-0.5 g/dL and superiority if the lower bound was ≥0 g/dL; p = 0.515, ANOVA — The p-value for hemoglobin change from Baseline (Day 1) was adjusted for baseline hemoglobin level and hemodialysis status; Treatment Difference = 0.10, 95% CI 2-sided [-0.21 to 0.41] — The 95% CI for hemoglobin change from Baseline (Day 1) was from an ANOVA model and adjusted for baseline hemoglobin level and hemodialysis status
Statistical Analysis 2: Comparison: Ferumoxytol vs Iron Sucrose; Without Imputation (Sensitivity Analysis): The p-value and two-sided 95% CI for the treatment difference in mean change in hemoglobin from Baseline (Day 1) to Week 5 were generated based on an ANOVA model adjusted for baseline hemoglobin level and hemodialysis status; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.587, ANOVA — [p-value comment as in outcome 1, analysis 1]; Treatment Difference = 0.09, 95% CI 2-sided [-0.23 to 0.41] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage Of Participants With An Increase In Hemoglobin ≥1.0 g/dL From Day 1 (Baseline) To Week 5
Description: The percentage of participants who achieved a ≥1.0 g/dL increase in hemoglobin at any time from Baseline (Day 1) up to Week 5 by treatment group is presented by study visit. Baseline hemoglobin for each participant was the Day 1 hemoglobin value (prior to injection of the study drug).
Time Frame: Baseline (Day 1) and up to Week 5
Population: ITT Population: Any randomized participant who had any exposure to study drug (IV ferumoxytol or IV iron sucrose).
Measure: Count of Participants; unit: Participants
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 80 | 82
Participants
  Week 2 | 20 | 11
  Week 3 | 32 | 20
  Week 4 | 37 | 31
  Week 5 | 40 | 34

ADVERSE EVENTS:
Arm/Group | Ferumoxytol | Iron Sucrose
Serious Adverse Events (participants affected / at risk) | 7/80 | 6/82
Other Adverse Events (participants affected / at risk) | 35/80 | 50/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferumoxytol (N=80) | Iron Sucrose (N=82)
Abscess limb (Infections and infestations) | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Peritoneal adhesions (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ferumoxytol (N=80) | Iron Sucrose (N=82)
Nasopharyngitis (Infections and infestations) | 3 | 2
Urinary tract infection (Infections and infestations) | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Injection site pain (General disorders) | 1 | 2
Edema peripheral (General disorders) | 2 | 6
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Headache (Nervous system disorders) | 3 | 2
Parosmia (Nervous system disorders) | 0 | 4
Hypotension (Vascular disorders) | 2 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Gout (Metabolism and nutrition disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Catheter site erythema (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 1
Injection site haematoma (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Device leakage (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Feeling cold (General disorders) | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal abscess (Infections and infestations) | 1 | 0
Urethritis (Infections and infestations) | 0 | 1
Burn first degree (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Facial palsy (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1
Treatment noncompliance (Social circumstances) | 0 | 1
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Poor veneous access (Vascular disorders) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data has been received by Sponsor, the Site and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.